CLINICAL TRIAL: NCT03572283
Title: Phase 1 Window of Opportunity Study of Parasympathetic Stimulation With Bethanechol in Localized Pancreatic Adenocarcinoma Prior to Surgery
Brief Title: Bethanechol Prior to Pancreatic Surgery
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Susan E. Bates, Professor of Medicine at Columbia University Medical Ctr, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AAAR6735
Record Dates: First submitted 2018-05-08; First posted 2018-06-28 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Pancreas Cancer
Keywords: Pancreas; pancreatic adenocarcinoma; adenocarcinoma; bethanechol; parasympathetic
MeSH Terms: conditions — Pancreatic Neoplasms; Adenocarcinoma | interventions — Bethanechol

STUDY DESIGN:
Intervention Model Description: Phase 0 study to assess the impact of bethanechol on pancreatic cancer biomarkers
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Bethanechol (Experimental): Patients with pancreatic adenocarcinoma will receive bethanechol prior to pancreatic surgery
  Interventions: Drug: Bethanechol

INTERVENTIONS:
Drug: Bethanechol — Supplied as 50mg oral tablets. Take 2 tablets (total 100mg) twice daily from day 1 for a minimum of 1 week and a maximum of 4 weeks (or 2 days prior to scheduled surgery). Medication should be taken 1 hour before meals in the morning and the evening. Although bethanechol is FDA approved, in this study its use is experimental.
  Other Names: Bethanechol chloride tablet

SUMMARY:
The primary objective of this study is to assess the impact of bethanechol therapy on tumor activity by looking at biomarkers of proliferation, inflammation, and stem cell markers in post-treatment specimens compared to pre-treatment specimens and compared to other patients who were not treated with bethanechol prior to surgery. The investigators hypothesize that treatment with bethanechol will alter nerve conduction within tumors by stimulating the parasympathetic nervous system and reduce tumor proliferation, reduce macrophage activation, reduce tumor necrosis factor (TNF) alpha, and decrease human cluster of differentiation 44 (CD44) protein cancer stem cells.

The safety objective is to assess the safety and tolerability of short course bethanechol prior to surgery and the impact of this treatment on immediate surgical outcomes. The investigators will assess all treatment-related toxicities with an emphasis on GI side effects and evaluate the impact of therapy on surgical delays or immediate post-op complications. All subjects will be contacted 1 week after beginning therapy to assess toxicity including GI specific toxicity and followed for safety for 30 days following completion of study medication. The investigators hypothesize that treatment for a minimum of 1 week will be tolerable in this selected patient population and will not interfere with progression to surgery or lead to increased surgical complications.

DETAILED DESCRIPTION:
Pancreatic ductal adenocarcinoma (PDA) is one of the most difficult cancers and, unlike other common cancers, annual deaths from PDA are rising. During the year 2017, it was estimated that 53,670 people would be diagnosed with PDA and approximately 43,090 people would die in the U.S. Despite recent advances, cytotoxic chemotherapy for PDA has been disappointing with response rates of 20-30% for the most active regimens and little activity for targeted therapies. Even among the small subset of patients who are suitable for surgical resection at the time of diagnosis, complete resection is followed by recurrence in >90% of patients without further systemic therapy, with a median time to recurrence of 6.9 months. Thus all PDA patients require systemic chemotherapy and more effective regimens are urgently needed.

The purpose of this study is to determine whether the drug, bethanechol, could potentially be used in combination with surgery to decrease the chance of cancer coming back after it is removed. Bethanechol is a medication that is approved by the FDA and regulates the parasympathetic nervous system. It is used to treat dry mouth and for patients who have difficulty urinating. It has been used to manage the side effects of chemotherapy drugs. The investigators planned this study in pancreatic cancer because animal models have shown that treatment with bethanechol can inhibit cancer growth and spread. People with pancreatic cancer localized to a small area usually undergo surgery to remove the tumor. The study is designed to investigate that the medication is easy to tolerate and that it shows signs of slowing cancer cell growth.

.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent for the trial.
* Age ≥18 years of age on the day of signing informed consent.
* Have histologically or cytologically confirmed the diagnosis of resectable pancreatic ductal adenocarcinoma or be willing to undergo a biopsy with confirmed pathology prior to starting therapy.
* Have a predicted life expectancy of greater than 3 months.
* Have a performance status of 0 or 1 using the Eastern Cooperative Oncology Group (ECOG) Performance Status Scale within 3 days of the first dose of study drug.
* Have a negative urine or serum pregnancy test within 7 days prior to receiving the first dose of study medication (Cycle 1, Day 1) (female subjects of childbearing potential). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required

Exclusion Criteria:

* Has received prior chemotherapy or radiotherapy for a current episode of pancreatic adenocarcinoma.
* Is currently using an acetylcholinesterase inhibitor or a beta-blocker.
* Has active peptic ulcer disease as defined by documented peptic ulcer and symptoms uncontrolled with oral medication.
* Has a known hypersensitivity or allergy to bethanechol.
* Has uncontrolled hyperthyroidism, defined as clinical hyperthyroidism uncontrolled by oral medication.
* Has bradycardia with resting heart rate < 50 beats per minute.
* Has chronic hypotension with resting systolic blood pressure < 90 mmHg.
* Has symptomatic coronary artery disease, such as angina or symptoms of claudication
* Has vasomotor instability.
* Has seizure disorder or required anti-seizure medication for seizure prevention within 5 years prior to study entry.
* Has a history of Parkinson's disease.
* Has bronchial asthma.
* Has a history of recent urinary bladder surgery within 12 months of study entry.
* Has a history of gastrointestinal resection and anastomosis within 12 months of study entry.
* Has a history of current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has a known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-04-08 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-08-24 (Actual)

PRIMARY OUTCOMES:
Change in cell proliferation by Ki-67 expression in tumor cells | Baseline, 28 days after surgery
  Individual tumor tissues will be evaluated, comparing pre-treatment and post-treatment samples. Percentage of change in proliferation/staining and standard deviation will be analyzed and calculated.

SECONDARY OUTCOMES:
Number of Adverse Events | Baseline, 28 days after surgery
  Subjects will be contacted every week (+/- 3 days) after the start of treatment to approximately 28 days after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Susan E Bates, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No